CLINICAL TRIAL: NCT01384474
Title: Impact of Crew Resource Management Training to Improve the Effectiveness of Surgical Safety Checklist
Brief Title: Impact of Crew Resource Management Training to Improve the Effectiveness of Surgical Safety Checklist (IDILIC)
Acronym: IDILIC
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50737; PHRC National 2010 (Other: government)
Record Dates: First submitted 2011-06-21; First posted 2011-06-29 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Surgery
Keywords: Crew Resource Management; Surgical safety checklist; Postoperative complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CRM training of surgical teams: CRM : Crew resource Management
  Interventions: Other: Diffusion of a surgical safety checklist
- No CRM training of surgical teams: CRM : Crew resource Management

INTERVENTIONS:
Other: Diffusion of a surgical safety checklist — * Assistance by a local caregiver investigator (i.e., surgeon, anaesthetist, nurse,...) responsible for the implementation of surgical safety checklist within the operatory rooms of his department ;
  * A two-step CRM training of surgical teams (i.e., surgeons, anaesthetists, nurses,...) conducted by advisors from the world of air company using video support:
    * First month following randomization: a course about the implementation of surgical safety checklist (using online-available WHO short movies and other videos of surgical teams) and core concepts of CRM adapted to the operating room;
    * Sixth month following randomization: a feedback to surgical teams aiming at identifying and solving barriers related to the checklist implementation and interpersonal communication
  * Written reminders including the systematic presence of an unfilled surgical safety checklist in the patient's medical report, stickers and wall posters in operatory rooms
  Groups: CRM training of surgical teams

SUMMARY:
This multicenter cluster-randomized trial will evaluate the impact of Crew Resource Management training on the occurrence of postoperative complications and the adherence to a surgical safety checklist, among a large sample of French surgical departments.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Hospitalization ≥ 24 hours
* Available medical file

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients needing a surgery who are hospitalized in one of the 31 departments.
Sampling Method: Non-Probability Sample
Enrollment: 23056 (Actual)
Dates: Start 2011-09; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of any major postoperative complication during hospitalization | during the two phases of the study : 18 months

SECONDARY OUTCOMES:
Team's adherence to the items of surgical safety checklist | During the two phases of the study : 18 months
Occurrence of any postoperative death during hospitalization | During the two phases of the study : 18 months
Healthcare workers' attitude regarding the patient safety culture | Twice during the study : the 4th and the 17th month after the beginning of the study

CONTACTS AND LOCATIONS:
Overall Officials: Cyrille COLIN, Principal Investigator — Hospices Civils de Lyon - Pôle Imer - 162 Avenue Lacassagne - 69003 LYON
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Sens F, Viprey M, Piriou V, Peix JL, Herquelot E, Occelli P, Bourdy S, Gawande AA, Carty Mj MJ, Michel P, Lifante JC, Colin C, Duclos A; IDILIC Study Group. Safety Attitude of Operating Room Personnel Associated With Accurate Completion of a Surgical Checklist: A Cross-sectional Observational Study. J Patient Saf. 2022 Aug 1;18(5):449-456. doi: 10.1097/PTS.0000000000000954. Epub 2021 Dec 17. PMID 35948294
- [Derived] Duclos A, Peix JL, Piriou V, Occelli P, Denis A, Bourdy S, Carty MJ, Gawande AA, Debouck F, Vacca C, Lifante JC, Colin C; IDILIC Study Group. Cluster randomized trial to evaluate the impact of team training on surgical outcomes. Br J Surg. 2016 Dec;103(13):1804-1814. doi: 10.1002/bjs.10295. Epub 2016 Sep 19. PMID 27642053